CLINICAL TRIAL: NCT00930657
Title: CO2 Inhalation and Risk for Panic Disorder
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090177; 09-M-0177
Record Dates: First submitted 2009-06-27; First posted 2009-06-30 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08-12

CONDITIONS: Panic Disorder
Keywords: Panic Disorder; Separation Anxiety; Familial; Risk; Respiratory Physiology
MeSH Terms: conditions — Panic Disorder; Anxiety, Separation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Objective:

To examine respiratory/physiological and subjective responding as well as genetic transmission among offspring of parents with a history of or current panic disorder (PD) diagnosis to determine whether diagnoses/symptoms, endophenotypes, or genetic profiles in offspring is differentially related to parent PD subtypes (i.e., respiratory and non-respiratory panic).

Study population:

Approximately 400 offspring of about 200 parents with current or past PD. Approximately 200 offsping/100 parents with PD will be enrolled at NIH/NIMH and the remainder at Virginia Commonwealth University in Richmond, VA.

Design:

A high-risk family design will be used wherein parents with either a current or past diagnosis of PD who have an offspring(s) (ages 9 to 20) will be recruited.

<TAB>

Outcome measures:

Outcome measures will include physiological recordings of respiratory, cardiac, and electrodermal responding during a 10 minute baseline followed by 15 minutes of 5% carbon dioxide enriched air (CO2). Research participants also will complete parent and child self-report measures and provide a DNA sample using a saliva protocol. A full listing of self-reports is provided in the Outcome Measures Section.

DETAILED DESCRIPTION:
Objective:

The objective of this study is to examine respiratory/physiological and subjective responding as well as genetic transmission among offspring of parents with a history of or current panic disorder (PD) diagnosis. Our goal is to determine whether diagnoses/symptoms, endophenotypes, or genetic profiles in offspring is differentially related to parent PD subtypes (i.e., respiratory and non-respiratory panic).

Study population:

Approximately 80 offspring between the ages of 9 and 20 years of age who have a parent with a current or past history of PD will be recruited. Approximately 40 offspring will be enrolled at NIH/NIMH and the remainder at Virginia Commonwealth University in Richmond, VA.

Design:

Offspring(s) between the ages of 9 to 20 who have a parent with a history of PD will be recruited. A complete psychiatric history will be obtained on all child participants. Child participants also will complete questionnaire measures, provide a sample of DNA, and participate in a carbon dioxide CO(2) lab challenge. The CO(2) lab challenge is the primary outcome measure.

Outcome measures:

Our primary outcome measures include physiological recordings of respiratory, cardiac, and electrodermal responding during a 10 minute baseline followed by 15 minutes of 5% carbon dioxide enriched air (CO(2). Research participants also will complete parent and child self-report measures and provide a DNA sample using a saliva protocol. A full listing of self-reports is provided in the Outcome Measures Section.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Children age 9-18, and young adults 18-20 who have a parent with a past or current history of PD.

EXCLUSION CRITERIA (ALL PARTICIPANTS):

* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease, one or more past seizures without a clear and resolved etiology,
* Subjects who are currently at high risk for homicide or suicide,
* Subjects with symptoms of psychosis
* Subjects with current DSM-IV substance abuse or dependence within the past year.
* Subjects with IQ<70,

ADDITIONAL EXCLUSION CRITERIA FOR CHILDREN:

* mania,
* pervasive developmental disorder,
* use of psychotropic medication,
* Child participants must be psychotropic free for at least 14 days prior to the CO(2) challenge session.
* For children taking fluoxetine, they must be free of this medication for at least 4 weeks.
* The proband parent must be a legal guardian of the child to qualify for the study.

Offspring passing screening criteria will be scheduled for an intake to complete a clinical interview, questionnaires, and CO(2) challenge task with assessment of respiratory physiology.

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-06-26; Study Completion 2019-08-12

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Abrams K, Rassovsky Y, Kushner MG. Evidence for respiratory and nonrespiratory subtypes in panic disorder. Depress Anxiety. 2006;23(8):474-81. doi: 10.1002/da.20179. PMID 16841338
- [Background] Battaglia M, Ogliari A, Harris J, Spatola CA, Pesenti-Gritti P, Reichborn-Kjennerud T, Torgersen S, Kringlen E, Tambs K. A genetic study of the acute anxious response to carbon dioxide stimulation in man. J Psychiatr Res. 2007 Dec;41(11):906-17. doi: 10.1016/j.jpsychires.2006.12.002. Epub 2007 Jan 24. PMID 17254605
- [Background] Biber B, Alkin T. Panic disorder subtypes: differential responses to CO2 challenge. Am J Psychiatry. 1999 May;156(5):739-44. doi: 10.1176/ajp.156.5.739. PMID 10327907